CLINICAL TRIAL: NCT07177742
Title: Prospective Cohort Study on the Relationship Between Peroxiredoxin 1 (PRDX1) in Blood Exosomes From Colorectal Cancer Radical Resection Specimens and Postoperative Liver Metastasis
Brief Title: Prospective Cohort Study on the Relationship Between Exosomal Peroxiredoxin 1 (PRDX1) and Postoperative Liver Metastasis
Status: Recruiting | Type: Observational
Sponsor: Mu-qing Yang (Other)
Responsible Party: Sponsor-Investigator, Mu-qing Yang, Associate Professor, Associate Attending Physician, Shanghai Tongji Hospital, Tongji University School of Medicine
Organization: Shanghai Tongji Hospital, Tongji University School of Medicine (Other)
Other Study IDs: K-2024-017
Record Dates: First submitted 2025-09-10; First posted 2025-09-17 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Colorectal Cancer; Liver Metastases From Colorectal Cancer; Pathology; Exosome; Peroxidized Redox Protein 1
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Specimens were retained in -80 ℃ refrigerator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- A surgical resectable colorectal cancer patients are set as prospective cohort.: The blood obtained from surgical resection specimens of resectable colorectal cancer patients was used to extract their serum exosomes and detect the concentration of PRDX1. The patients were aged 19-80 years and were planned to be included in a prospective follow-up cohort of 252. The occurrence of metastasis was observed, and the predicted and critical values of PRDX1 concentration in portal vein branch serum exosomes obtained from the specimens were analyzed.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Observation.

SUMMARY:
The occurrence of liver metastasis after curative surgery for resectable colorectal cancer is an important cause of death for patients. Accurately identifying high-risk patients for metastasis and intervening in them has important clinical significance. The pathological examination of surgical specimens failed to fully utilize valuable specimen information and accurately predict liver metastasis; The biomarkers secreted by tumors are metabolized in the liver through the portal vein, especially the particles such as extracellular vesicles secreted by tumors, which are ultimately diluted in peripheral blood and cannot be effectively detected. Our research group extracted an average of 11.25ml of blood (named blood derived from portal vein branch specimens, sdBlood for short) from 8 colorectal cancer radical surgery specimens. Compared with peripheral blood, protein mass spectrometry analysis revealed a significant increase in exosome proteins such as peroxidized redox protein 1 (PRDX1), which are highly correlated with metastasis. This project innovatively uses sdBlood, which has been overlooked by routine pathological examination, to detect the exosomal protein PRDX1 in sdBlood, which is significantly higher than the peripheral blood concentration. A prospective cohort study was established, including 252 patients with pathologically confirmed colorectal cancer after radical surgery. The incidence and time of liver metastasis were followed up and observed. Cox regression statistical analysis was used to determine the correlation between this marker and metastasis and determine its critical value, providing a basis for clinical diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 19-80 years old, gender not limited;

  * Can comply with the requirements of the research visit plan and other protocols;

    * Voluntarily participate and sign an informed consent form; ④ Diagnosed with colon adenocarcinoma through pathological examination; ⑤ Patients who have completed colorectal radical surgery.

Exclusion Criteria:

* Patients who cannot complete radical surgery for colorectal cancer;

  * Patients with liver diseases (chronic hepatitis B, hepatitis C, severe fatty liver, cirrhosis);

    * Patients who require combined organ resection;

      * Combine patients with other malignant tumors or blood or immune system diseases; ⑤ Prior to tumor resection, any anti-tumor treatment, including radiotherapy, chemotherapy, and molecular targeted therapy, has been performed; ⑥ After surgery, it was found that the mesenteric vein branch of the specimen could not obtain blood due to severe infiltration or other reasons.

        * Patients with severe postoperative complications leading to delayed treatment (Clavien-Dindo grade III or above).

Ages: 19 Months to 80 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Local resectable colorectal cancer patients aged 19-80 years who have not undergone preoperative radiotherapy or chemotherapy and have no distant metastasis.
Sampling Method: Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2021-02-15 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Liver metastasis. | From enrollment to 5 years after coloretal radical surgery.
  During the follow-up period, the study subjects exhibited liver metastatic lesions (at least on nodal with enhanced and diameter over 1 cm, or diameter over 0.5cm with increased diameter during consecutive two followups) on imaging examinations (enhanced abdominal CT, enhanced MRI, or 18FDP-PET scan), which were confirmed as liver metastasis after interpretation by a deputy chief surgeon and a physician with a position higher than deputy chief in radiology.

SECONDARY OUTCOMES:
Local recurrence. | From enrollment to 5 years after colorectal radical resection.
  During the follow-up period, the study subjects exhibited local lesions over 1cm on imaging examinations (enhanced abdominal CT, enhanced MRI, or 18FDP-PET scan), which were confirmed as liver metastasis after interpretation by a deputy chief surgeon and a physician with a position higher than deputy chief in radiology. During the follow-up period, the study subjects exhibited liver metastatic lesions on imaging examinations (enhanced abdominal CT, enhanced MRI, or 18FDP-PET scan), which were confirmed as local recurrence after interpretation by a deputy chief surgeon and a physician with a position higher than deputy chief in radiology.
Lung metastasis. | From enrollment to 5 years after colorectal radical resection.
  During the follow-up period, the study subjects exhibited new lesions (at least on nodal with enhanced and diameter over 1 cm, or diameter over 0.5cm with increased diameter during consecutive two followups) on imaging examinations (chest plain CT, or 18FDP-PET scan), which were confirmed as lung metastasis after interpretation by a deputy chief surgeon and a physician with a position higher than deputy chief in radiology.
Peritoneal recurrence. | From enrollment to 5 years after colorectal radical resection.
  During the follow-up period, the study subjects exhibited new peritoneal lesions (at least on nodal with enhanced and diameter over 1 cm, or diameter over 0.5cm with increased diameter during consecutive two followups) on imaging examinations (enhanced abdominal CT, enhanced MRI, or 18FDP-PET scan), which were confirmed as peritoneal metastasis after interpretation by a deputy chief surgeon and a physician with a position higher than deputy chief in radiology.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Tongji Hospital, Hepatobilliary Surgery Center, Tongji University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided